CLINICAL TRIAL: NCT01648829
Title: Pharmacodynamic Comparison of Pitavastatin Versus Atorvastatin on Platelet Reactivity in Patients With Coronary Artery Disease Treated With Dual Antiplatelet Therapy - The PORTO Trial
Brief Title: PharmacOdynamic compaRison of piTavastatin Versus atOrvastatin on Platelet Reactivity
Acronym: PORTO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 449/2012/D
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): os, 20 mg, once per day, for 30 days
  Interventions: Drug: Atorvastatin
- Pitavastatin (Active Comparator): os, 4 mg, once per day, for 30 days
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Atorvastatin — Patients will receive randomly atorvastatin (20 mg day) for 30 days
  Other Names: Torvast, Pfizer, USA
  Arms: Atorvastatin
Drug: Pitavastatin — Patients will receive randomly pitavastatin (4 mg day) for 30 days
  Other Names: Livalo, Kowa Pharmaceuticals, Japan
  Arms: Pitavastatin

SUMMARY:
Levels of platelet reactivity in patients on Dual Antiplatelet Therapy (DAPT) can be influenced by concomitant treatment with medications (i.e. statins) that inhibit the CYP3A4 system involved in the activation of clopidogrel. Atorvastatin and simvastatin are metabolized by CYP3A4. Pitavastatin, unlike other statins, is little metabolized, most of the dose being excreted unchanged in bile, and biotransformation through the cytochrome P450 system is minimal. Indeed, pitavastatin's cyclopropyl group diverts the drug away from metabolism by CYP3A4 and allows only a small amount of clinically insignificant metabolism by CYP2C9.

The primary objective of this study is to compare the pharmacodynamic effects of a CYP3A4-metabolized statin (atorvastatin) versus a non-CYP3A4-metabolized statin (pitavastatin) in patients showing high platelet reactivity while on DAPT.

DETAILED DESCRIPTION:
Patients with coronary artery disease (CAD) are often treated with dual anti-platelet therapy (DAPT), including aspirin and clopidogrel, to prevent from recurrent atherothrombotic events.

Levels of platelet reactivity in patients on DAPT can be influenced by concomitant treatment with medications (i.e. statins) that inhibit the CYP3A4 system involved in the activation of clopidogrel.

Atorvastatin and simvastatin are metabolized by CYP3A4. Pitavastatin, unlike other statins, is little metabolized, most of the dose being excreted unchanged in bile, and biotransformation through the cytochrome P450 system is minimal. Indeed, pitavastatin's cyclopropyl group diverts the drug away from metabolism by CYP3A4 and allows only a small amount of clinically insignificant metabolism by CYP2C9.

At least 1 month after starting DAT (clopidogrel 75 mg and aspirin 100 mg), patients will receive randomly atorvastatin (20 mg day, N=50) or pitavastatin (4 mg day, N=50) for 30 days (until T-1).

At this time-point, there will be a wash-out period of 15 days after the first treatment with atorvastatin or pitavastatin in order to avoid any carry-over effect.

Afterwards, a cross-over will be performed, and patients will be switched to the other drug which will be continued for further 30 days (until T-2).

No previous studies have evaluated the influence of pitavastatin as compared with other statins on platelet reactivity in patients receiving DAPT.

The primary objective of this study is to compare the pharmacodynamic effects of a CYP3A4-metabolized statin (atorvastatin) versus a non-CYP3A4-metabolized statin (pitavastatin) in patients showing high platelet reactivity while on DAPT.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Class I indication to DAT because of recent (< 12 months) percutaneous coronary intervention and/or recent acute coronary syndrome (< 12 months)
* Stable clinical conditions
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

* Use of other drug interfering with CYP activity such as proton pump inhibitors
* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 30 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California])

SECONDARY OUTCOMES:
Frequency of high platelet reactivity | After 30 days of treatment with each drug
  Frequency of high platelet reactivity with the 2 study treatments (as defined by a Platelet Reaction Unit value>208)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University, Rome, Italy